CLINICAL TRIAL: NCT03053050
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of Selonsertib in Subjects With Nonalcoholic Steatohepatitis (NASH) and Bridging (F3) Fibrosis
Brief Title: Safety and Efficacy of Selonsertib in Adults With Nonalcoholic Steatohepatitis (NASH) and Bridging (F3) Fibrosis
Acronym: STELLAR-3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated early due to lack of efficacy based on the results of the Week 48 analysis as prespecified in the clinical study protocol.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-384-1943; 2016-004374-18 (EudraCT Number)
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Results first posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — selonsertib

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SEL 18 mg (Experimental): Randomized Phase: Selonsertib (SEL) 18 mg tablet + placebo to match SEL 6 mg tablet for 240 weeks
  Open-Label (OL) Phase: Participants who experience a hepatic clinical event or have biopsy confirmed progression to cirrhosis during the randomized phase, prior to completing the Week 240 visit, will be offered the option to roll over into an OL phase to receive OL SEL 18 mg for a total treatment duration of 240 weeks inclusive of the randomized phase.
  Interventions: Drug: SEL; Drug: Placebo to match SEL 6 mg
- SEL 6 mg (Experimental): Randomized Phase: SEL 6 mg tablet + placebo to match SEL 18 mg tablet for 240 weeks
  OL Phase: Participants who experience a hepatic clinical event or have biopsy confirmed progression to cirrhosis during the randomized phase, prior to completing the Week 240 visit, will be offered the option to roll over into an OL phase to receive OL SEL 18 mg for a total treatment duration of 240 weeks inclusive of the randomized phase.
  Interventions: Drug: SEL; Drug: Placebo to match SEL 18 mg
- Placebo (Placebo Comparator): Randomized Phase: Placebo to match SEL 6 mg tablet + placebo to match SEL 18 mg tablet for 240 weeks
  OL Phase: Participants who experience a hepatic clinical event or have biopsy confirmed progression to cirrhosis during the randomized phase, prior to completing the Week 240 visit, will be offered the option to roll over into an OL phase to receive OL SEL 18 mg for a total treatment duration of 240 weeks inclusive of the randomized phase.
  Interventions: Drug: Placebo to match SEL 6 mg; Drug: Placebo to match SEL 18 mg

INTERVENTIONS:
Drug: SEL — Tablets administered orally once daily
  Other Names: selonsertib; GS-4997
  Arms: SEL 18 mg; SEL 6 mg
Drug: Placebo to match SEL 6 mg — Tablets administered orally once daily
  Arms: Placebo; SEL 18 mg
Drug: Placebo to match SEL 18 mg — Tablets administered orally once daily
  Arms: Placebo; SEL 6 mg

SUMMARY:
The primary objective of this study is to evaluate whether selonsertib (SEL; GS-4997) can cause fibrosis regression and reduce progression to cirrhosis and associated complications in adults with NASH and bridging (F3) fibrosis.

ELIGIBILITY:
Key Inclusion Criteria:

* Liver biopsy consistent with NASH and bridging (F3 fibrosis) according to the NASH Clinical Research Network (CRN) classification in the opinion of the central reader
* Has the following laboratory parameters at the screening visit:

  * Alanine aminotransferase (ALT) ≤ 8 x upper limit of normal (ULN)
  * Creatinine Clearance (CLcr) ≥ 30 milliliter/minute (mL/min), as calculated by the Cockcroft-Gault equation
  * Hemoglobin A1c (HbA1c) ≤ 9.5% (or serum fructosamine ≤ 381 μmol if HbA1c is unable to be resulted)
  * Total bilirubin ≤ 1.3 x ULN (unless an alternate etiology such as Gilbert's syndrome or hemolytic anemia is present)

Key Exclusion Criteria:

* Prior history of decompensated liver disease including clinical ascites, hepatic encephalopathy (HE), or variceal bleeding
* Child-Pugh (CP) score > 6, as determined at screening, unless due to therapeutic anti-coagulation
* Model for End-stage Liver Disease (MELD) score > 12, as determined at screening, unless due to therapeutic anti-coagulation
* Other causes of liver disease including, but not limited to, alcoholic liver disease, hepatitis B, hepatitis C, autoimmune disorders, drug-induced hepatotoxicity, Wilson disease, iron overload, and alpha-1-antitryspin deficiency, based on medical history and/ or centralized review of liver histology.
* History of liver transplantation
* Current or history of hepatocellular carcinoma (HCC)

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 808 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (298):
- United States (124):
  - Institute of Liver Health, Chandler, Arizona
  - Banner University Medical Center-Phoenix, Phoenix, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Baptist Medical Center, Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - eStudySite, Chula Vista, California
  - Southern California Liver Centers, Coronado, California
  - United Gastroenterologists, Costa Mesa, California
  - TriWest Research Associates, LLC, El Cajon, California
  - Fresno Clinical Research Center, Fresno, California
  - University of California San Diego (UCSD), La Jolla, California
  - Ruane Clinical Research Group, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - eStudySite, Oceanside, California
  - California Liver Institute, Pasadena, California
  - Inland Empire Liver Foundation, Rialto, California
  - University of California, Davis Medical Center, Sacramento, California
  - Medical Associates Research Group, San Diego, California
  - Kaiser Permanente, San Diego, California
  - California Pacific Medical Center - Sutter Pacific Medical Foundation San Francisco Center for Liver Disease Dept. of Transplant, San Francisco, California
  - Mission Gastroenterology and Hepatology, San Francisco, California
  - University of California San Francisco (UCSF), San Francisco, California
  - Silicon Valley Research Institute, San Jose, California
  - University of Colorado, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Integrity Clinical Research, LLC, Doral, Florida
  - UF Hepatology Research at CTRB, Gainesville, Florida
  - UF Health Jacksonville-Gastroenterology Emerson, Jacksonville, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - Sunrise Medical Research, Inc, Lauderdale Lakes, Florida
  - Sunrise Research Institute, Miami, Florida
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - Genoma Research Group, Inc, Miami, Florida
  - Advanced Research Institute, New Port Richey, Florida
  - Avail Clinical Research, LLC, Orange City, Florida
  - South Florida Center of Gastroenterology, PA, Wellington, Florida
  - Florida Medical Clinic, PA, Zephyrhills, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Piedmont Transplant Institute, Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Northwestern Memorial Hospital; Clinical Research Unit, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - NorthShore University Healthsystem, Glenview, Illinois
  - Indiana University Health - University Hospital, Indianapolis, Indiana
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Gastroenterology Associates of Hazard, Hazard, Kentucky
  - Delta Research Partners, LLC, Bastrop, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ocshner Medical Center, New Orleans, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Digestive Disease Associates, PA, Catonsville, Maryland
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Gastroenterology Associates of Western Michigan, P.L.C., Wyoming, Michigan
  - Huron Gastroenterology Associates/Center for Digestive Care, Ypsilanti, Michigan
  - University of Minnesota Medical Center - Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Southern Therapy and Advanced Research LLC (STAR), Ridgeland, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Kansas City Gastroenterology and Hepatology, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - eStudySite, Las Vegas, Nevada
  - Rutgers New Jersey Medical School- Doctors Office Center, Newark, New Jersey
  - University of Buffalo, Clinical and Translational Research Center, Buffalo, New York
  - Northwell Health - Sandra Atlas Bass Center for Liver Diseases, Manhasset, New York
  - Icahn School of Medicine at Mount Sinai Beth Israel, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill / UNC School of Medicine, Chapel Hill, North Carolina
  - Duke University Medical Center - Duke South Clinics, Durham, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Triad Clinical Trials LLC, Greensboro, North Carolina
  - Piedmont HealthCare, d/b/a Carolinas Center for Liver Disease, Huntersville, North Carolina
  - PMG Research of Rocky Mount, LLC, Rocky Mount, North Carolina
  - Piedmont HealthCare, d/b/a Carolinas Center for Liver Disease, Statesville, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - UC Health/Holmes Hospital, Cincinnati, Ohio
  - Northeast Clinical Research Center, LLC, Bethlehem, Pennsylvania
  - Hospital of the University of Pennsylvania- Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC - Center for Liver Diseases at the Thomas E. Starlz Institute, Pittsburgh, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - eStudySite, Pittsburgh, Pennsylvania
  - Guthrie Medical Group, PC, Sayre, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System - Gastroenterology and Liver Center, Greenville, South Carolina
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Gastro One, Germantown, Tennessee
  - Quality Medical Research PLLC, Nashville, Tennessee
  - Vanderbilt University Medical Center - Digestive Disease Center, Nashville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Pinnacle Clinical Research, PLLC, Austin, Texas
  - Austin Center for Clinical Research, Austin, Texas
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Texas Digestive Disease Consultants, Dallas, Texas
  - Baylor Scott & White All Saints Medical Center, Fort Worth, Texas
  - Kelsey-Seybold Clinic, Houston, Texas
  - Baylor College of Medicine - Advanced Liver Therapies, Houston, Texas
  - VAMC & Baylor College, Houston, Texas
  - Pinnacle Clinical Research, PLLC, Live Oak, Texas
  - American Research Corporation, The Texas Liver Institute, San Antonio, Texas
  - Intermountain Liver Disease and Transplant Center, Murray, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - The University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Verity Research, Inc., Fairfax, Virginia
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Emeritas Research Group, Lansdowne Town Center, Virginia
  - Bon Secours St. Mary's Hospital of Richmond, Inc. d/b/a Bon Secours Liver Institute of Virginia, Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Bon Secours St. Mary's Hospital of Richmond, Inc. d/b/a Bon Secours Liver Institute of Virginia, Richmond, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Virginia Mason, Seattle, Washington
  - Swedish Organ Transplant and Liver Center, Seattle, Washington
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
- Argentina (2):
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Instituto Oulton, Córdoba
- Australia (10):
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - St. George's Hospital, Kogarah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Health, Monash Medical Centre, Clayton, Victoria
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - The Alfred Hospital, Alfred Health, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Austria (2):
  - Medizinische Universitat Graz, Universitatsklinik fue Innere Medizin, Graz
  - Allgemeines Krankenhaus Wien, Vienna
- Belgium (3):
  - CUB Hopital Erasme, Brussels
  - UZ Brussel, Brussels
  - Universitaire Ziekenhuizen Leuven, Leuven
- Brazil (5):
  - Hospital das Clínicas da Faculdade de Medicina de Botucatu - FMB/Universidade Estadual Paulista Julio de Mesquita Filho - UNESP, Botucatu
  - Hospital de Clínicas de Porto Alegre - HCPA/UFRGS, Porto Alegre
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto - USP, Ribeirão Preto
  - Hospital Das Clinicas Da Faculdade De Medicina Da Universidade De Sao Paulo, São Paulo
  - Universidade Federal de São Paulo / Unidade Ambulatorial de Pesquisa Clínica - I (UAPC-I), São Paulo
- Canada (11):
  - University of Calgary Liver Unit (Heritage Medical Research Clinic), Calgary, Alberta
  - University of Alberta Hospital - Walter C. Mackenzie Health Sciences Centre (WMC), Edmonton, Alberta
  - LAIR Centre, Vancouver, British Columbia
  - Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - (G.I.R.I.) GI Research Institute, Vancouver, British Columbia
  - PerCuro Clinical Research Ltd., Victoria, British Columbia
  - South Shore Medical Arts, Bridgewater, Nova Scotia
  - William Osler Health System-Brampton Civic Hospital, Brampton, Ontario
  - South Shore Medical Arts, London, Ontario
  - Toronto Center for Liver Diseases (TCLD), Toronto General Hospital, Toronto, Ontario
  - Chronic Viral Illness Service/Royal Victoria Hospital/McGill University Health Centre (MUHC), Montreal, Quebec
- France (15):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Centre Hospitalier Universitaire Estaing, Clermont-Ferrand
  - Hopital Henri Mondor, Créteil
  - CHU de Grenoble- Hopital Michallon, Grenoble
  - Centre Hospitalier Regional Universitaire- Hopital Claude Huriez, Lille
  - CHU de Limoges- Hopital Dupuytren- Federation Hepatologie, Limoges
  - Hopital de la Croix Rousse, Lyon
  - Hôpital Saint Joseph, Marseille
  - Centre Hospitalier Universitaire de Nice- Hopital l'Archet 2, Nice
  - Hopital Cochin, Paris
  - Hopital Beaujon, Pessac
  - Centre Hospitalier Universitaire de Bordeaux, Pessac
  - Centre Hospitalier Universitaire de Strasbourg- Nouvel Hopital Civil, Strasbourg
  - Centre Hospitalier Universitaire de Toulouse- Hopital Purpan, Toulouse
  - Hopital Paul Brousse, Villejuif
- Germany (9):
  - Uniklinik RWTH Aachen, Medizinische Klinik III, Aachen
  - Zentrum fur Infektiologie Berlin Prenzlauer Berg GmbH (zibp), Berlin
  - Universitatsklinikum Bonn (AoR), Bonn
  - Universitatsklinikum Frankfurt der Goethe-Universitat, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Uniklinikum des Saarlandes- Klinik fur Innere Medizin II, Homburg
  - Gastroenterologisch- Hepatologisches Zentrum Kiel, Kiel
  - Eugastro Gmbh, Leipzig
  - Johannes Gutenberg-Universitat, Mainz
- Hong Kong (2):
  - Alice Ho Miu Ling Nethersole Hospital, Tai Po
  - Tuen Mun Hospital, Tuenmen
- India (8):
  - Midas Multispecialty Hospital, Nagpur, Maharashtra
  - Institute of Post Graduate Medical Education and Research / SSKM Hospital, Kolkata
  - Kasturba Medical College (KMC) Hospital, Mangalore
  - Global Hospital-Super Speciality & Transplant Centre (A Unit of Centre for Digestive and Kidney Diseases (India) Pvt. Ltd.), Mumbai
  - Maharaja Agrasen Hospital, New Delhi
  - All India Institute of Medical Sciences, New Delhi
  - Fortis Flt. Lt. Rajan Dhall Hospital, New Delhi
  - Institute of Liver & Biliary Sciences, New Delhi
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - The Lady Davis Carmel Medical Center, Haifa
  - Holy Family hospital, Nazareth
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (3):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - IRCCS Ospedale Casa Sollievo Della Soferrenza, San Giovanni Rotondo
- Japan (37):
  - Chiba University Hospital, Chiba
  - Fukui-Ken Saiseikai Hospital, Fukui-shi
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - Tokyo Medical University Ibaraki Medical Center, Ibaraki
  - Juntendo University Shizuoka Hospital, Izunokuni
  - Kagoshima University Medical And Dental Hospital, Kagoshima
  - Kanazawa University Hospital, Kanagawa
  - Nara Medical University Hospital, Kashihara
  - Toranomon Hospital Kajigaya, Kawasaki
  - Shinkokura Hospital, Kitakyushu
  - Kumamoto Shinto General Hospital, Kumamoto
  - Kurume University Hospital, Kurume
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Shinshu University Hospital, Matsumoto
  - Toranomon Hospital, Minato
  - Miyazaki Medical Center Hospital, Miyazaki
  - Japanese Red Cross Musashino Hospital, Musashino
  - Aichi Medical University Hospital, Nagakute
  - Heart Life Hospital, Nakagami
  - Nara City Hospital, Nara
  - Hyogo College of Medicine Hospital, Nishinomiya
  - Kawasaki Medical School General Medical Center, Okayama
  - Okayama University Hospital, Okayama
  - National Hospital Organization Osaka National Hospital, Osaka
  - National Hospital Organization Nagasaki Medical Center, Ōmura
  - Hirakata Kohsai Hospital, Ōsaka
  - Saga University Hospital, Saga
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital, Sapporo
  - Tohoku Rosai Hospital, Sendai
  - National Center for Global Health and Medicine Hospital, Shinjuku-ku
  - Saiseikai Suita Hospital, Suita
  - Kagawa Prefectural Central Hospital, Takamatsu
  - Ehime University Hospital, Tōno
  - Mie University Hospital, Tsu
  - Yamagata University Hospital, Yamagata
  - Yokohama City University Hospital, Yokohama
- Malaysia (2):
  - Hospital Selayang, Batu Caves
  - University of Malaya Medical Centre, Kuala Lumpur
- Mexico (3):
  - Phylasis Clinicas Research S. de RL de CV., Cuautitlán
  - Consultorio Médico, Mexico City
  - Investigaciones Medicas Cisneros SC, Monterrey
- University Medical Center Utrecht, Utrecht, Netherlands
- Auckland City Hospital, Grafton, New Zealand
- Poland (2):
  - Szpital Specjalistyczny Nr 1 w Bytomiu, Oddzial Obserwacyjno-Zakazny i Hepatologii, Bytom
  - Wojewodzki Specjalistyczny Szpital im. W. Bieganskiego, Lodz
- Centro Hospitalar de Tras-os-Montes e Alto Douro, E.P.E, Vila Real, Portugal
- Puerto Rico (3):
  - Klinical Investigations Group, LLC, San Juan
  - VA Caribbean Healthcare System, San Juan
  - Fundacion de Investigacion de Diego, San Juan
- Singapore (5):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital Pte Ltd., Singapore
  - Khoo Teck Puat Hospital, Singapore
- South Korea (11):
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - National Health Insurance Service- Ilsan Hospital, Goyang-si
  - Hanyang University Seoul Hospital, Seoul
  - Asan Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (9):
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Puerto de Hierro Majadahonda, Majadahonda
  - CHOP_Complejo Hospitalrio Universitario de Pontevedra, Pontevedra
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Switzerland (2):
  - Universitätsklinik für Viszerale Chirurgie und Medizin, Inselspital, Hepatologie, Bern
  - Istituto Cantonale di Patologia Locarno, Lugano
- Taiwan (12):
  - Changhua Christian Hospital, Chang-hua
  - Ditmanson Medical Foundation Chia-Yi Christian Hospital, Chiayi City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-DA Hospital, Kaohsiung City
  - Chang Gung Medical Foundation, Keelung Chang Gung Memorial Hospital, Keelung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospitalv, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Cathay General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation, Linkou Chang Gung Memorial Hospital, Taoyuan District
- United Kingdom (10):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Derby Teaching Hospitals NHS FT, Derby
  - University Hospitals Birmingham NHS Foundation Trust, Edgbaston
  - King's College Hospital NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Portsmouth Hospitals NHS Trust, Portsmouth
  - Abertawe Bro Morgannwg University Health Board, Swansea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Anstee QM, Lawitz EJ, Alkhouri N, Wong VW, Romero-Gomez M, Okanoue T, Trauner M, Kersey K, Li G, Han L, Jia C, Wang L, Chen G, Subramanian GM, Myers RP, Djedjos CS, Kohli A, Bzowej N, Younes Z, Sarin S, Shiffman ML, Harrison SA, Afdhal NH, Goodman Z, Younossi ZM. Noninvasive Tests Accurately Identify Advanced Fibrosis due to NASH: Baseline Data From the STELLAR Trials. Hepatology. 2019 Nov;70(5):1521-1530. doi: 10.1002/hep.30842. Epub 2019 Aug 19. PMID 31271665
- [Result] Alkhouri N, Younossi ZM, Lawitz EJ, Wong VWS, Romero-Gomez M, et al. Impact of age on routinely available noninvasive tests for the discrimination of advanced fibrosis due to NASH in the phase 3 STELLAR trials of the ASK1 inhibitor selonsertib [Poster SAT-273]. European Association for the Study of the Liver (EASL); 2019; Vienna Austria.
- [Result] Younossi ZM, Stepanova M, Anstee QM, Lawitz EJ, Wai-Sun Wong V, Romero-Gomez M, Kersey K, Li G, Subramanian GM, Myers RP, Djedjos CS, Okanoue T, Trauner M, Goodman Z, Harrison SA. Reduced Patient-Reported Outcome Scores Associate With Level of Fibrosis in Patients With Nonalcoholic Steatohepatitis. Clin Gastroenterol Hepatol. 2019 Nov;17(12):2552-2560.e10. doi: 10.1016/j.cgh.2019.02.024. Epub 2019 Feb 16. PMID 30779990
- [Result] Anstee QM, Lawitz EJ, Alkhouri N, Wai Sun Wong V, Romero-Gomez M, et al. Routinely available noninvasive tests discriminate advanced fibrosis due to NASH in the Phase 3 STELLAR trials of the ASK1 inhibitor selonsertib [poster]. American Association for the Study of Liver Diseases (AASLD); 2018, San Francisco, CA.
- [Result] Younossi ZM, Lawitz E, Alkhouri N, Wong VWS, Romero-Gomez M, et al. Algorithms using noninvasive tests can accurately identify patients with advanced fibrosis due to NASH: Data From the STELLAR clinical trials [Poster LB-10]. AASLD; 2018; San Francisco, CA.
- [Result] Younossi ZM, Stepanova M, Anstee QM, Lawitz EJ, Wai-Sun Wong V, et al. Severe impairment of patient-reported outcomes in patients with advanced fibrosis due to non-alcoholic steatohepatitis (NASH) [Poster]. AASLD; 2018; San Francisco, CA.
- [Result] Younossi ZM, Stepanova M, Anstee QM, Lawitz EJ, Wai Sun Wong V, et al. Advanced fibrosis based on noninvasive tests in nonalcoholic steatohepatitis (NASH) is associated with impairment of patient-reported outcomes [Poster]. AASLD; 2018; San Francisco, CA.
- [Derived] Loomba R, Huang DQ, Sanyal AJ, Anstee QM, Trauner M, Lawitz EJ, Ding D, Ma L, Jia C, Billin A, Huss RS, Chung C, Goodman Z, Wong VW, Okanoue T, Romero-Gomez M, Abdelmalek MF, Muir A, Afdhal N, Bosch J, Harrison S, Younossi ZM, Myers RP. Liver stiffness thresholds to predict disease progression and clinical outcomes in bridging fibrosis and cirrhosis. Gut. 2023 Mar;72(3):581-589. doi: 10.1136/gutjnl-2022-327777. Epub 2022 Sep 9. PMID 36750244
- [Derived] Younossi ZM, Anstee QM, Wai-Sun Wong V, Trauner M, Lawitz EJ, Harrison SA, Camargo M, Kersey K, Subramanian GM, Myers RP, Stepanova M. The Association of Histologic and Noninvasive Tests With Adverse Clinical and Patient-Reported Outcomes in Patients With Advanced Fibrosis Due to Nonalcoholic Steatohepatitis. Gastroenterology. 2021 Apr;160(5):1608-1619.e13. doi: 10.1053/j.gastro.2020.12.003. Epub 2020 Dec 8. PMID 33307033
- [Derived] Harrison SA, Wong VW, Okanoue T, Bzowej N, Vuppalanchi R, Younes Z, Kohli A, Sarin S, Caldwell SH, Alkhouri N, Shiffman ML, Camargo M, Li G, Kersey K, Jia C, Zhu Y, Djedjos CS, Subramanian GM, Myers RP, Gunn N, Sheikh A, Anstee QM, Romero-Gomez M, Trauner M, Goodman Z, Lawitz EJ, Younossi Z; STELLAR-3; STELLAR-4 Investigators. Selonsertib for patients with bridging fibrosis or compensated cirrhosis due to NASH: Results from randomized phase III STELLAR trials. J Hepatol. 2020 Jul;73(1):26-39. doi: 10.1016/j.jhep.2020.02.027. Epub 2020 Mar 6. PMID 32147362
- [Derived] Younossi ZM, Stepanova M, Younossi I, Racila A. Validation of Chronic Liver Disease Questionnaire for Nonalcoholic Steatohepatitis in Patients With Biopsy-Proven Nonalcoholic Steatohepatitis. Clin Gastroenterol Hepatol. 2019 Sep;17(10):2093-2100.e3. doi: 10.1016/j.cgh.2019.01.001. Epub 2019 Jan 11. PMID 30639779

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Asia, Europe, Australia, South America, Puerto Rico, and New Zealand. The first participant was screened on 13 February 2017. The last study visit occurred on 19 June 2019.
Pre-assignment Details: 2250 participants were screened.
Groups:
- SEL 18 mg: Randomized Phase: Selonsertib (SEL) 18 mg tablet orally once daily + placebo to match SEL 6 mg tablet orally once daily for 240 weeks.
- SEL 6 mg: Randomized Phase: SEL 6 mg tablet orally once daily + placebo to match SEL 18 mg tablet orally once daily for 240 weeks.
- Placebo: Randomized Phase: Placebo-to-match SEL 6 mg tablet orally once daily + placebo to match SEL 18 mg tablet orally once daily for 240 weeks.
- Open-Label SEL 18 mg: Open-Label (OL) Phase: Participants who experienced a hepatic clinical event or have biopsy confirmed progression to cirrhosis during the randomized phase, prior to completing the Week 240 visit, were offered the option to roll over into an OL phase to receive OL SEL 18 mg daily for a total treatment duration of 240 weeks inclusive of the randomized phase.
Period: Randomized Phase
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo | Open-Label SEL 18 mg
Started | 324 | 323 | 161 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 324 | 323 | 161 | 0
Not completed — Study Terminated by Sponsor | 259 | 260 | 128 | 0
Not completed — Withdrew Consent | 16 | 8 | 9 | 0
Not completed — Investigator's Discretion | 6 | 6 | 3 | 0
Not completed — Lost to Follow-up | 5 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Randomized but Never Treated | 2 | 2 | 2 | 0
Not completed — Entered the Open-Label Phase | 36 | 45 | 18 | 0
Period: Open-label Phase
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo | Open-Label SEL 18 mg
Started | 0 | 0 | 0 | 99 (Participants with hepatic clinical event or progression to cirrhosis had option to go into OL Phase.)
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 99
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 89
Not completed — Withdrew Consent | 0 | 0 | 0 | 6
Not completed — Investigator's Discretion | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- SEL 18 mg: Randomized Phase: Selonsertib (SEL) 18 mg tablet orally once daily + placebo to match SEL 6 mg tablet orally once daily for 240 weeks
  Open-Label (OL) Phase: Participants who experienced a hepatic clinical event or have biopsy confirmed progression to cirrhosis during the randomized phase, prior to completing the Week 240 visit, were offered the option to roll over into an OL phase to receive OL SEL 18 mg daily for a total treatment duration of 240 weeks inclusive of the randomized phase.
- SEL 6 mg: Randomized Phase: SEL 6 mg tablet orally once daily + placebo to match SEL 18 mg tablet orally once daily for 240 weeks
  OL Phase: Participants who experienced a hepatic clinical event or have biopsy confirmed progression to cirrhosis during the randomized phase, prior to completing the Week 240 visit, were offered the option to roll over into an OL phase to receive OL SEL 18 mg daily for a total treatment duration of 240 weeks inclusive of the randomized phase.
- Placebo: Randomized Phase: Placebo to match SEL 6 mg tablet orally once daily + placebo to match SEL 18 mg tablet orally once daily for 240 weeks
  OL Phase: Participants who experienced a hepatic clinical event or have biopsy confirmed progression to cirrhosis during the randomized phase, prior to completing the Week 240 visit, were offered the option to roll over into an OL phase to receive OL SEL 18 mg daily for a total treatment duration of 240 weeks inclusive of the randomized phase.
- Total: Total of all reporting groups
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo | Total
Number analyzed (Participants) | 322 | 321 | 159 | 802
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (9.1) | 57 (9.2) | 57 (9.0) | 57 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181 | 196 | 76 | 453
  Male | 141 | 125 | 83 | 349
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = Local regulators did not allow collection of race or ethnicity information.
  Participants
    Race: American Indian or Alaska Native | 5 | 1 | 2 | 8
    Race: Asian | 88 | 84 | 41 | 213
    Race: Black | 8 | 5 | 2 | 15
    Race: White | 219 | 227 | 113 | 559
    Race: Other | 2 | 3 | 1 | 6
    Race: Not Permitted | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = Local regulators did not allow collection of race or ethnicity information.
  Participants
    Ethnicity: Not Hispanic or Latino | 269 | 269 | 137 | 675
    Ethnicity: Hispanic or Latino | 52 | 48 | 22 | 122
    Ethnicity: Not Permitted | 1 | 4 | 0 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 161 | 172 | 80 | 413
  Japan | 38 | 23 | 19 | 80
  Canada | 16 | 14 | 8 | 38
  France | 14 | 10 | 5 | 29
  South Korea | 8 | 13 | 7 | 28
  Australia | 9 | 12 | 3 | 24
  Hong Kong | 10 | 8 | 6 | 24
  Spain | 9 | 10 | 4 | 23
  Taiwan | 7 | 14 | 0 | 21
  United Kingdom | 8 | 5 | 7 | 20
  India | 7 | 4 | 4 | 15
  Germany | 4 | 3 | 4 | 11
  Singapore | 4 | 5 | 2 | 11
  Brazil | 3 | 4 | 2 | 9
  Israel | 2 | 4 | 3 | 9
  Belgium | 3 | 3 | 2 | 8
  Mexico | 5 | 2 | 1 | 8
  Italy | 2 | 4 | 0 | 6
  Argentina | 3 | 2 | 0 | 5
  Austria | 2 | 2 | 0 | 4
  Poland | 2 | 2 | 0 | 4
  Puerto Rico | 2 | 1 | 0 | 3
  Switzerland | 1 | 0 | 2 | 3
  Malaysia | 1 | 1 | 0 | 2
  Portugal | 0 | 2 | 0 | 2
  Netherlands | 0 | 1 | 0 | 1
  New Zealand | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a ≥ 1-Stage Improvement in Fibrosis According to the Nonalcoholic Steatohepatitis (NASH) Clinical Research Network (CRN) Classification Without Worsening of NASH at Week 48
Description: Fibrosis improvement was defined as ≥ 1-stage decrease from baseline in fibrosis according to the NASH CRN classification. NASH CRN fibrosis stages range from 0 to 4, with higher scores indicating greater fibrosis (0=None, 4=Cirrhosis). Worsening of NASH was defined as ≥ 1 point increase from baseline in hepatocellular ballooning or lobular inflammation according to the Non-Alcoholic Fatty Liver Disease (NAFLD) Activity Score (NAS) criteria. As defined by NAS, hepatocellular ballooning ranges from 0-2 and lobular inflammation ranges from 0-3, with higher scores indicating more severe hepatocellular ballooning or lobular inflammation.
Time Frame: Week 48
Population: The Full Analysis Set included all participants who were randomized into the study and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo
Number analyzed (Participants) | 322 | 321 | 159
percentage of participants | 9.6 [6.6 to 13.4] | 12.1 [8.8 to 16.2] | 13.2 [8.4 to 19.5]
Statistical Analysis 1: Comparison: SEL 18 mg vs Placebo; Test type: Superiority; p = 0.4941, Mantel Haenszel — Difference between SEL 18 mg and Placebo, 95% confidence interval (CI) and p-value were obtained by stratum-adjusted Mantel-Haenszel method with baseline diabetes mellitus status and Enhanced Liver Fibrosis (ELF) test score as stratification factors; Percentage Difference = -2.1, 95% CI 2-sided [-8.3 to 4.0]
Statistical Analysis 2: Comparison: SEL 6 mg vs Placebo; Test type: Superiority; p = 0.9321, Mantel Haenszel — Difference between SEL 6 mg and Placebo, 95% CI and p-value were obtained by stratum-adjusted Mantel-Haenszel method with baseline diabetes mellitus status and ELF test score as stratification factors; Percentage Difference = -0.3, 95% CI 2-sided [-6.6 to 6.0]

2. Primary Outcome: Event-Free Survival (EFS) at Week 240 as Assessed by Time to First Clinical Event
Description: EFS was assessed by the time to the first clinical event, including progression to cirrhosis on liver biopsy, liver decompensation events, liver transplantation, and all-cause mortality.
Time Frame: Week 240
Population: No data was analyzed as the study was terminated and no participants reached the Week 240 timepoint.
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants Who Had Progression to Cirrhosis at Week 48
Description: Progression to cirrhosis was defined as a change in NASH CRN fibrosis stage from < 4 at baseline to 4 at Week 48.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo
Number analyzed (Participants) | 322 | 321 | 159
percentage of participants | 13.0 [9.6 to 17.2] | 15.6 [11.8 to 20.0] | 15.7 [10.4 to 22.3]
Statistical Analysis 1: Comparison: SEL 18 mg vs Placebo; Test type: Superiority; p = 0.2593, Mantel Haenszel — Difference between SEL 18 mg and Placebo, 95% CI and p-value were obtained by stratum-adjusted Mantel-Haenszel method with baseline diabetes mellitus status and ELF test score as stratification factors; Percentage Difference = -4.0, 95% CI 2-sided [-10.8 to 2.9]
Statistical Analysis 2: Comparison: SEL 6 mg vs Placebo; Test type: Superiority; p = 0.8080, Mantel Haenszel — Difference between SEL 6 mg vs Placebo, 95% CI and p-value were obtained by stratum-adjusted Mantel-Haenszel method with baseline diabetes mellitus status and ELF test score as stratification factors; Percentage Difference = -0.9, 95% CI 2-sided [-7.9 to 6.1]

4. Secondary Outcome: Percentage of Participants Who Had a ≥ 1-Stage Improvement in Fibrosis Without Worsening of NASH at Week 240
Description: Fibrosis improvement was defined as ≥ 1-stage decrease from baseline in fibrosis according to the NASH CRN classification. NASH CRN fibrosis stages range from 0 to 4, with higher scores indicating greater fibrosis (0=None, 4=Cirrhosis). Worsening of NASH was defined as ≥ 1 point increase from baseline in hepatocellular ballooning or lobular inflammation according to the NAS criteria. As defined by NAS, hepatocellular ballooning ranges from 0-2 and lobular inflammation ranges from 0-3, with higher scores indicating more severe hepatocellular ballooning or lobular inflammation.
Time Frame: Week 240
Population: No data was analyzed as the study was terminated and no participants reached the Week 240 timepoint.
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants Who Had a ≥ 1-Stage Improvement in Fibrosis at Week 48
Description: Fibrosis improvement was defined as ≥ 1-stage decrease from baseline in fibrosis according to the NASH CRN classification. NASH CRN fibrosis stages range from 0 to 4, with higher scores indicating greater fibrosis (0=None, 4=Cirrhosis).
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo
Number analyzed (Participants) | 322 | 321 | 159
percentage of participants | 12.7 [9.3 to 16.9] | 13.7 [10.1 to 18.0] | 16.4 [11.0 to 23.0]
Statistical Analysis 1: Comparison: SEL 18 mg vs Placebo; Test type: Superiority; p = 0.5636, Mantel Haenszel — [p-value comment as in outcome 3, analysis 1]; Percentage Difference = -2.0, 95% CI 2-sided [-8.7 to 4.8]
Statistical Analysis 2: Comparison: SEL 6 mg vs Placebo; Test type: Superiority; p = 0.5915, Mantel Haenszel — [p-value comment as in outcome 1, analysis 2]; Percentage Difference = -1.9, 95% CI 2-sided [-8.6 to 4.9]

6. Secondary Outcome: Percentage of Participants Who Had a ≥ 1-Stage Improvement in Fibrosis at Week 240
Description: as for outcome 5
Time Frame: Week 240
Population: No data was analyzed as the study was terminated and no participants reached the Week 240 timepoint.
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants Who Had NASH Resolution Without Worsening of Fibrosis at Week 48
Description: NASH resolution was defined as lobular inflammation of 0 or 1 from ≥ 1 at baseline and hepatocellular ballooning of 1 from a value ≥ 1 at baseline; both criteria were necessary conditions. Evaluable participants had baseline lobular inflammation and hepatocellular ballooning ≥ 1. Worsening of Fibrosis was defined by an increase in Fibrosis stage from 3 to 4 as defined by NASH CRN.
Time Frame: Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo
Number analyzed (Participants) | 322 | 321 | 158
percentage of participants | 5.0 [2.9 to 7.9] | 4.4 [2.4 to 7.2] | 8.9 [4.9 to 14.4]
Statistical Analysis 1: Comparison: SEL 18 mg vs Placebo; Test type: Superiority; p = 0.2455, Mantel Haenszel — [p-value comment as in outcome 3, analysis 1]; Percentage Difference = -3.2, 95% CI 2-sided [-8.5 to 2.2]
Statistical Analysis 2: Comparison: SEL 6 mg vs Placebo; Test type: Superiority; p = 0.1371, Mantel Haenszel — [p-value comment as in outcome 1, analysis 2]; Percentage Difference = -4.0, 95% CI 2-sided [-9.3 to 1.3]

8. Secondary Outcome: Percentage of Participants Who Had NASH Resolution Without Worsening of Fibrosis at Week 240
Description: as for outcome 7
Time Frame: Week 240
Population: No data was analyzed as the study was terminated and no participants reached the Week 240 timepoint.
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose date up to last dose (maximum: 111.4 weeks) plus 30 days
Description: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Placebo: Randomized Phase: Placebo to match SEL 6 mg tablet orally once daily + placebo to match SEL 18 mg tablet orally once daily for 240 weeks.
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo | Open-Label SEL 18 mg
All-Cause Mortality (participants affected / at risk) | 0/322 | 0/321 | 0/159 | 0/99
Serious Adverse Events (participants affected / at risk) | 47/322 | 36/321 | 17/159 | 6/99
Other Adverse Events (participants affected / at risk) | 248/322 | 254/321 | 130/159 | 48/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SEL 18 mg (N=322) | SEL 6 mg (N=321) | Placebo (N=159) | Open-Label SEL 18 mg (N=99)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Internal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis relapsing (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis of male external genital organ (Infections and infestations) | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 0 | 0
Postoperative abscess (Infections and infestations) | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 2 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 2 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Pancreatic leak (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ammonia increased (Investigations) | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastatic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 1 | 0
Schizoaffective disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 0
Cystitis interstitial (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Testicular necrosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hepatic hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SEL 18 mg (N=322) | SEL 6 mg (N=321) | Placebo (N=159) | Open-Label SEL 18 mg (N=99)
Abdominal distension (Gastrointestinal disorders) | 13 | 12 | 8 | 2
Abdominal pain (Gastrointestinal disorders) | 22 | 27 | 15 | 3
Abdominal pain upper (Gastrointestinal disorders) | 33 | 26 | 16 | 5
Constipation (Gastrointestinal disorders) | 40 | 43 | 19 | 4
Diarrhoea (Gastrointestinal disorders) | 52 | 47 | 30 | 8
Nausea (Gastrointestinal disorders) | 32 | 39 | 14 | 6
Vomiting (Gastrointestinal disorders) | 19 | 18 | 8 | 1
Fatigue (General disorders) | 35 | 33 | 12 | 3
Oedema peripheral (General disorders) | 18 | 9 | 4 | 3
Hepatic cirrhosis (Hepatobiliary disorders) | 42 | 50 | 25 | 0
Bronchitis (Infections and infestations) | 23 | 21 | 6 | 1
Influenza (Infections and infestations) | 19 | 20 | 14 | 4
Nasopharyngitis (Infections and infestations) | 46 | 40 | 21 | 0
Sinusitis (Infections and infestations) | 21 | 21 | 12 | 5
Upper respiratory tract infection (Infections and infestations) | 41 | 46 | 21 | 6
Urinary tract infection (Infections and infestations) | 14 | 27 | 13 | 3
Contusion (Injury, poisoning and procedural complications) | 10 | 5 | 8 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 | 30 | 18 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 33 | 27 | 11 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 | 17 | 7 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 | 18 | 8 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 15 | 11 | 5
Dizziness (Nervous system disorders) | 16 | 30 | 2 | 2
Headache (Nervous system disorders) | 36 | 38 | 18 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 18 | 14 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 23 | 20 | 11 | 3

LIMITATIONS AND CAVEATS:
Based on the results of the Week 48 analysis, the study was terminated early for lack of efficacy as prespecified in the clinical study protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/50/NCT03053050/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/50/NCT03053050/SAP_001.pdf